CLINICAL TRIAL: NCT04195958
Title: A Multicenter, Open-Label, Single-Arm Study to Assess the Impact of Omalizumab on Exercise Capacity, Physical Activity, and Sleep Quality in Patients With Moderate to Severe Allergic Asthma
Brief Title: A Study to Assess the Impact of Omalizumab on Exercise Capacity, Physical Activity, and Sleep Quality in Participants With Moderate to Severe Allergic Asthma
Acronym: EDURO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to low enrollment, this study was terminated early.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML41615
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Moderate-to-severe Allergic Asthma
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omalizumab (Experimental)
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Omalizumab will be administered by subcutaneous (SC) injection at a dose of 150 milligrams (mg) to 375 mg every 2 or 4 weeks. The dose and frequency will be determined by body weight (kg) and the level of total IgE (IU/mL) measured during screening.

SUMMARY:
This study will assess the effect of omalizumab on exercise capacity, physical activity, and sleep quality after 24 weeks of treatment in participants with moderate to severe allergic asthma. Exercise capacity will be assessed using cardiopulmonary exercise testing (CPET). Physical activity and sleep quality will be assessed with a wearable physical activity and sleep monitor. The study will consist of a 4-week screening period, a 24-week treatment period, and a 4-week safety follow-up. Approximately 60 participants will be enrolled, and omalizumab will be dosed according to the approved United States Package Insert (USPI) dosing table.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma for at least 12 months prior to screening
* Documented history of positive skin test or in vitro reactivity to a perennial aeroallergen
* Able to comply with asthma control medication adherence, digital monitoring data collection, and eDiary requirements during screening period
* Able to safely complete incremental exercise tolerance at screening
* Pre-bronchodilator FEV1 of 40%-80% of predicted at screening
* Documented history of variable airflow obstruction or hyper-responsiveness within 12 months of study entry
* On inhaled corticosteroids (ICS) therapy at a total daily dose greater than or equal to (≥)500 micrograms (ug) of fluticasone propionate or equivalent and at least one second controller (LABA, LAMA, LTRA) for ≥3 months prior to screening
* Uncontrolled asthma during the screening period, defined as an ACQ-5 ≥0.75 score
* Sleep disturbance due to asthma (e.g. cough, wheezing etc.) in the opinion of the investigator
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or to use adequate contraception during the treatment period and for 60 days after the final dose of study drug.

Exclusion Criteria:

* Known history of anaphylaxis/hypersensitivity to omalizumab
* Treatment with investigational drugs within 12 weeks or 5 half-lives (whichever is longer) prior to screening
* Treatment with monoclonal antibodies (e.g., omalizumab, mepolizumab, dupilumab) for 6 months prior to screening
* Maintenance oral corticosteroid therapy, defined as daily or alternate-day oral corticosteroid within 3 months prior to screening or during the screening period
* Treatment with systemic (oral, IV, or IM) corticosteroids within 4 weeks prior to screening or during the screening period
* Isolated diagnosis of exercise induced asthma without chronic symptoms
* History of interstitial lung disease, COPD, or other clinically significant lung disease other than asthma
* Current malignancy or history of malignancy within 5 years prior to screening
* Unable to complete cardiopulmonary exercise testing and/or perform physical activity due to underlying cardiac, neurologic or orthopedic conditions
* Ongoing physician-treated sleep disorder that is unrelated to asthma within 6 months prior to screening
* Current smoker or past smoker with >10 pack years
* Known HIV infection at screening
* Known acute or chronic infections with hepatitis C virus (HCV) and hepatitis B virus (HBV) at screening
* Infection that resulted in hospital admission, required treatment with intravenous or intramuscular antibiotics within 4 weeks prior to screening, or any active infection that required treatment with oral antibiotics within 2 weeks prior to screening
* Active tuberculosis requiring treatment within 12 months prior to screening
* History of alcohol, drug, or chemical abuse within 6 months of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (12):
- United States (12):
  - Peninsula Research Associates, Rolling Hills Estates, California
  - National Jewish Health, Denver, Colorado
  - Broward Research Center, Pembroke Pines, Florida
  - University of Iowa Hospitals & Clinics; Internal Medicine, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Lenox Hill Hospital, New York, New York
  - American Health Research Inc., Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Temple Uni Medical Center; Pulmonary & Critical Care Medicine, Philadelphia, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Swedish Health Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated by the Sponsor. Only 3 participants were enrolled in this study.
Groups:
- Omalizumab: Omalizumab was administered by subcutaneous (SC) injection at a dose of 150 milligrams (mg) to 375 mg every 2 or 4 weeks. The dose and frequency was determined by body weight (kg) and the level of total IgE (IU/mL) measured during screening.
Period: Overall Study
Arm/Group | Omalizumab
Started | 3
Completed | 1
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: This study was terminated by the Sponsor. Only 3 participants were enrolled in this study. Based on the low enrolment number and in order to protect and maintain participant privacy/confidentiality, no data is reported.
Arm/Group | Omalizumab
Number analyzed (Participants) | 0
Age, Continuous [unit: Years]
Sex: Female, Male
Race/Ethnicity, Customized

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 24 in Endurance Time (Minutes) During Cardiopulmonary Exercise Testing (CPET) at a Constant Work Rate (CWR)
Description: This study was terminated by the Sponsor. Only 3 participants were enrolled in this study. Based on the low enrolment number and in order to protect and maintain participant privacy/confidentiality, no data is reported.
Time Frame: From Baseline to Week 24
Population: as for baseline characteristics
Arm/Group | Omalizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline at Week 24 in Physical Activity (Minutes/Day) as Assessed by a Wearable Physical Activity and Sleep Monitor
Description: as for outcome 1
Time Frame: From Baseline to Week 24
Population: as for baseline characteristics
Arm/Group | Omalizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline at Week 24 in Dynamic Hyperinflation at Isotime, as Measured by Inspiratory Capacity During CPET at a CWR
Description: as for outcome 1
Time Frame: From Baseline to Week 24
Population: as for baseline characteristics
Arm/Group | Omalizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline at Week 24 in Sleep Efficiency as Assessed by a Wearable Physical Activity and Sleep Monitor
Description: as for outcome 1
Time Frame: From Baseline to Week 24
Population: as for baseline characteristics
Arm/Group | Omalizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Participants With Adverse Events
Description: as for outcome 1
Time Frame: From Baseline to Week 28
Population: as for baseline characteristics
Arm/Group | Omalizumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants With Serious Adverse Events
Description: as for outcome 1
Time Frame: From Baseline to Week 28
Population: as for baseline characteristics
Arm/Group | Omalizumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Participants With Adverse Events Leading to Discontinuation of Omalizumab
Description: as for outcome 1
Time Frame: From Baseline to Week 24
Population: as for baseline characteristics
Arm/Group | Omalizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Baseline to Week 28
Description: AEs were collected at each participant contact. Severity of AEs was assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Arm/Group | Omalizumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (N=3)
General Disorders (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was terminated by the Sponsor. Only 3 participants were enrolled in this study. Based on this, there were not enough participants enrolled to perform a meaningful analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT04195958/Prot_SAP_000.pdf